CLINICAL TRIAL: NCT02618512
Title: A Phase I/II Open Label Study in Previously Studied, SBC-103 Treatment Naïve MPS IIIB Subjects to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics/Efficacy of SBC-103 Administered Intravenously
Brief Title: A Open Label Study in Previously Studied, SBC-103 Treatment Naïve MPS IIIB Subjects to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics/Efficacy of SBC-103 Administered Intravenously
Acronym: CL01-T
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor's decision to terminate the SBC-103 program was reached after review of the data from all interventional clinical studies of SBC-103.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGLU-CL01-T; 2015-001983-20 (EudraCT Number)
Record Dates: First submitted 2015-10-21; First posted 2015-12-01 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Mucopolysaccharidosis III, Type B (MPS IIIB); Sanfilippo B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- SBC-103 (Experimental): Patients were administered 1 mg/kg by IV infusion once every other week (qow) for at least 12 weeks. After evaluation of 12-week safety, tolerability, and pharmacodynamic data in individual patients, the dose was increased to 3 mg/kg qow. Infusions were to be at least 10 days apart and were administered every 14 days ±5 days.
  Interventions: Drug: SBC-103

INTERVENTIONS:
Drug: SBC-103 — SBC-103 is a recombinant human alpha-N-acetylglucosaminidase (rhNAGLU). Patients were started with low dose of SBC-103 for 12 weeks and then will escalate to a higher dose.

SUMMARY:
This study evaluated the safety and tolerability of intravenous (IV) administration of SBC-103 in previously studied, SBC-103 treatment naïve patients with mucopolysaccharidosis III, type B (MPS IIIB, Sanfilippo B) who participated in the NGLU-CL01 study. The NGLU-CL01 study was a non-interventional study that evaluated structural brain abnormalities and blood brain barrier (BBB) integrity by magnetic resonance imaging (MRI) and cerebrospinal fluid/serum albumin index.

ELIGIBILITY:
Participants from NGU-CL01 study were enrolled into the NGLU-CL01-T study. Subjects who met all of the inclusion criteria and none of the exclusion criteria were eligible to participate in this study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SBC-103
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SBC-103
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of SBC-103
Description: The planned primary endpoint of this study was safety and tolerability of SBC-103 in patients with MPS IIIB, as measured by Number of participants with treatment-emergent adverse events, including serious adverse events; infusion-associated reactions; incidence of antidrug antibodies, clinical laboratory tests, cerebrospinal fluid findings, vital signs, and prior and concomitant medications
Time Frame: Planned duration was baseline to 164 weeks but due to early termination of the study, actual is 96 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | SBC-103
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Baseline to 96 Weeks.
Description: Treatment-emergent AEs by System Organ Class (SOC) and Preferred Term are classified according to the Medical Dictionary for Regulatory Activities (MedDRA) v19.0.
Arm/Group | SBC-103
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBC-103 (N=3)
Device Related Infection (Infections and infestations) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Catheter placement (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBC-103 (N=3)
Fall (Injury, poisoning and procedural complications) | 3 (8)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Pyrexia (General disorders) | 2 (5)
Gait disturbance (General disorders) | 1 (2)
Pain (General disorders) | 1 (2)
Complication associated with device (General disorders) | 1 (1)
Excessive granulation tissue (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (8)
Toothache (Gastrointestinal disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Vomiting projectile (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (11)
Staphylococcal infection (Infections and infestations) | 1 (2)
Candida infection (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Catheter site pain (General disorders) | 1 (2)
Restlessness (Psychiatric disorders) | 2 (4)
Anxiety (Psychiatric disorders) | 2 (3)
Sleep disorder (Psychiatric disorders) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Breath holding (Psychiatric disorders) | 1 (1)
Emotional distress (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Psychomotor hyperactivity (Nervous system disorders) | 2 (2)
Dyskinesia (Nervous system disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (2)
Motor dysfunction (Nervous system disorders) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1)
Skin warm (Skin and subcutaneous tissue disorders) | 2 (2)
Application site erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Hair disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Premenstrual pain (Reproductive system and breast disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Precocious puberty (Endocrine disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Body temperature increased (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early termination of the study only safety data are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Informed Consent Form (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02618512/ICF_000.pdf
  • Study Protocol (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT02618512/Prot_001.pdf
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT02618512/SAP_002.pdf